CLINICAL TRIAL: NCT04850690
Title: Effect of Cognitive and Motor Tasks on Gait in Individuals With Cerebral Palsy
Brief Title: Cognitive and Motor Tasks in Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, mbudak, Miray Budak, Istanbul Medipol University Hospital
Other Study IDs: CogMo-CP2021
Record Dates: First submitted 2021-04-14; First posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Cerebral Palsy; Gait Disorders, Neurologic; Cognitive Orientation; Motor Activity
Keywords: Cerebral Palsy; Cognitive Task; Dual Task Paradigm; Motor Task; Gait
MeSH Terms: conditions — Cerebral Palsy; Gait Disorders, Neurologic; Orientation, Spatial; Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with hemiparetic Cerebral palsy: 15 children with CP, between 9-15 years old
  Interventions: Diagnostic Test: 2D Gait analysis

INTERVENTIONS:
Diagnostic Test: 2D Gait analysis — The gait with four different conditions (single gait, Cognitive Task, Motor Task and Cognitive Task&Motor Task) was evaluated by Kinovea video analysis method on a 10-meter course.
  * Single: Walking without task at a self-selected speed
  * Cognitive Task (CT): Walking while counting down rhythmically from 20 in threes
  * Motor Task (MT): Walking while carrying an empty box
  * CT + MT: Walking while carrying an empty box and counting down rhythmically from 20 in threes

SUMMARY:
Various gait deviations are observed in children with cerebral palsy. Our aim was to determine the effect of cognitive task (CT) and motor task (MT) on gait in children with cerebral palsy (CP). 15 children with CP, between 9-15 years old, with Communication Function Classification System (CFSS) level I, with Gross Motor Function Classification System (GMFCS) and Manual Ability Classification System (MACS) level I-II were included in the study. The gait with four different conditions (single gait, CT, MT and CT&MT) was evaluated by Kinovea video analysis method on a 10-meter course.

Results:

DETAILED DESCRIPTION:
All children with CP were instructed to walk on the track under four different conditions:

* Single: Walking without task at a self-selected speed
* Cognitive Task (CT): Walking while counting down rhythmically from 20 in threes
* Motor Task (MT): Walking while carrying an empty box
* CT + MT: Walking while carrying an empty box and counting down rhythmically from 20 in threes

The task was explained to individuals by a physiotherapist. The individuals were not allowed to use orthosis during walking performance. Running was not accepted. 30 seconds were given to take a break between tasks. The physiotherapist followed the individuals along the track in case of any falling. If the child was not able to complete the track (falling or need to rest), the evaluation was accepted uncomplete and was excluded from the database.

The Kinovea-08.15 software program was used to assess all of the outputs (images and videos) from the camera

ELIGIBILITY:
Inclusion Criteria:

* having been diagnosed with CP in the health committee
* being between 9-15 years of age, having a mental level as "normal" (in terms of compliance with the exercises)
* being in Gross Motor Function Classification System (GMFSC) Level I-II
* being in Manual Ability Classification System (MACS) Level I-II
* being in Communication Function Classification System (CFSS) Level I (communication method is speech).

Exclusion Criteria:

* having a mental retardation
* having severe vision impairment
* underwenting Botulinum Toxin (BOTOX) injection or surgery affecting lower extremities in the last 6 months.

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 15 children with Cerebral Palsy, between 9-15 years old
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
2D Gait analysis | through study completion, an average of 1 year
  Kinovea video analysis

CONTACTS AND LOCATIONS:
Overall Officials: Miray BUDAK, PhD, Study Director — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided